CLINICAL TRIAL: NCT07187284
Title: Evaluating Endervascular Denervation (EDN) Combined With Transarterial Intervention (TACE/HAIC) and Second-Line Immune-Targeted Therapy in Locally Advanced Hepatocellular Carcinoma (HCC) With Portal Vein Tumor Thrombosis After Progression on First-Line Systemic Therapy: A Prospective, Multicenter, Randomized Controlled Study
Brief Title: EDN Combined With TACE/HAIC and Second-Line Immune-Targeted Treatment Versus TACE/HAIC Alone in Locally Advanced HCC With Portal Vein Tumor Thrombosis After First-Line Therapy Failure: A Prospective, Multicenter, Randomized Controlled Trial
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Dr. Teng was elected as an Academician of the Chinese Academy of Sciences in 2021 and as a Fellow of the Chinese Academy of Medical Sciences in 2022., Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZDSYLL382-P01
Record Dates: First submitted 2025-09-19; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: HCC - Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment intervention group (Experimental): Participants randomized to the treatment intervention group will receive the following combination therapy: 1.A single procedure of Endovascular Denervation (EDN): Percutaneous catheter-based ablation of the peri-arterial sympathetic nerves. 2.On-demand Transarterial Interventional Therapy: This consists of either Transarterial Chemoembolization (TACE) or Hepatic Arterial Infusion Chemotherapy (HAIC), administered based on individual patient's disease assessment and treatment response. 3.Second-line Immuno-Targeted Drug Therapy: Standard systemic therapy with a combination of immune checkpoint inhibitors and targeted agents (e.g., anti-PD-1/PD-L1 antibodies plus tyrosine kinase inhibitors or VEGF inhibitors). The specific drugs are not limited by the protocol and are chosen at the investigator's discretion according to local standards of care.
  Interventions: Combination Product: EDN combined with TACE/HAIC and Immuno-Targeted Therapy
- Control group (Active Comparator): Participants randomized to the control group will receive the current standard of care for the studied patient population, which consists of:
  1. On-demand Transarterial Interventional Therapy: This consists of either Transarterial Chemoembolization (TACE) or Hepatic Arterial Infusion Chemotherapy (HAIC), administered based on individual patient's disease assessment and treatment response.
  2. Second-line Immuno-Targeted Drug Therapy: Standard systemic therapy with a combination of immune checkpoint inhibitors and targeted agents (e.g., anti-PD-1/PD-L1 antibodies plus tyrosine kinase inhibitors or VEGF inhibitors). The specific drugs are not limited by the protocol and are chosen at the investigator's discretion according to local standards of care.
  Interventions: Combination Product: TACE/HAIC plus Immuno-Targeted Therapy

INTERVENTIONS:
Combination Product: EDN combined with TACE/HAIC and Immuno-Targeted Therapy — Experimental Intervention (Treatment Group):
  This arm evaluates a novel combination strategy. Participants will undergo a single session of Endovascular Denervation (EDN) in conjunction with standard care. The complete intervention includes:
  Endovascular Denervation (EDN): A one-time, catheter-based percutaneous procedure for the ablation of peri-arterial sympathetic nerves surrounding the common hepatic artery and/or proper hepatic artery. The procedure utilizes a multi-electrode radiofrequency ablation system (e.g., Netrod®). Ablation parameters are set to 60°C for 120 seconds per site, with a minimum of 20 ablations performed to ensure adequate denervation.
  On-demand Transarterial Intervention: Following EDN, participants will receive either Transarterial Chemoembolization (TACE) or Hepatic Arterial Infusion Chemotherapy (HAIC), as determined by the treating investigator based on individual patient anatomy and tumor characteristics.
  Arms: Treatment intervention group
Combination Product: TACE/HAIC plus Immuno-Targeted Therapy — This is the active comparator intervention representing the current standard-of-care regimen for the study population. Participants randomized to the control group will receive a combination of locoregional and systemic therapy, specifically excluding the experimental Endovascular Denervation (EDN) procedure.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of combining endovascular denervation (EDN) with transarterial chemoembolization/ hepatic arterial infusion chemotherapy (TACE/HAIC) plus second-line immune-targeted therapy in patients with locally advanced hepatocellular carcinoma (HCC) who have progressed after first-line systemic therapy and present with portal vein tumor thrombus (PVTT).

The main questions this study aims to answer are:

Does the addition of EDN to standard TACE/HAIC and immune-targeted therapy improve intrahepatic progression-free survival (hPFS) based on RECIST 1.1 criteria? What is the safety profile of the combined treatment, including device-related adverse events? Researchers will compare the experimental group (EDN + TACE/HAIC + immune-targeted therapy) with the control group (TACE/HAIC + immune-targeted therapy alone) in a 1:1 randomized design. A total of 62 participants will be enrolled across 8 centers, with an expected enrollment period of 12 months and a 12-month follow-up period.

Participants will:

Undergo screening assessments including imaging (CT/MRI), blood tests, and ECG within specified time windows.

Receive assigned interventions (EDN procedure or control) during the baseline visit (Day 0).

Attend follow-up visits at 1 month (±7 days), 3 months (±14 days), 6 months (±30 days), 9 months (±30 days), and 12 months (±30 days) for repeated imaging, laboratory tests, and safety evaluations.

Have their tumor response, survival outcomes, and adverse events monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years (inclusive), regardless of gender.
2. Diagnosis of CNLC Stage IIIa HCC with portal vein tumor thrombus (vp type 1-3) confirmed by histopathology, cytology, or imaging.
3. Progression of disease after first-line systemic therapy.
4. At least one measurable lesion according to RECIST 1.1 criteria.
5. Child-Pugh class A or B.
6. ECOG performance status of 0 to 2.
7. Scheduled to undergo TACE or HAIC treatment.
8. Adequate hematological, hepatic, and renal function within 14 days prior to study initiation, defined as:

White blood cell count ≥2.0×10⁹/L AND neutrophil count ≥1.0×10⁹/L. Platelet count ≥60×10⁹/L. Hemoglobin concentration ≥90 g/L. Total bilirubin ≤2.0 × upper limit of normal (ULN). Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5 × ULN. Albumin ≥2.8 g/dL. International normalized ratio (INR) ≤1.6. Creatinine ≤1.5 × ULN AND calculated creatinine clearance ≥30 mL/min.

Exclusion Criteria:

1. Preoperative abdominal CT or MR enhanced scan suggests celiac trunk anatomy is unsuitable for EDN procedure.
2. History of orthostatic hypotension.
3. Diffuse liver tumors or extensive extrahepatic metastases with an expected survival of <3 months.
4. Cachexia or multi-organ failure.
5. Severe hepatic dysfunction (Child-Pugh class C).
6. Uncorrectable coagulation dysfunction.
7. Presence of severe concurrent infection.
8. Accompanied by Vp4 type portal vein tumor thrombus.
9. Abnormal blood supply to the target lesion that precludes transarterial interventional therapy.
10. History of bilioenteric anastomosis within the past year.
11. Severe allergy to known contrast agents or embolization materials.
12. Pregnant or lactating women, or individuals with childbearing potential planning pregnancy during the trial period.
13. Clinically significant (e.g., active) cardiovascular disease, including:

    Unstable angina within ≤6 months prior to randomization. New York Heart Association (NYHA) class ≥II congestive heart failure. Poorly controlled arrhythmia despite medication (patients with controlled atrial fibrillation are eligible), or any clinically significant abnormality found on resting ECG.

    ≥Grade 3 peripheral vascular disease (e.g., symptomatic and interfering with activities of daily living, requiring intervention).

    Transient ischemic attack or subarachnoid hemorrhage within 6 months prior to randomization, or participation in other drug or device clinical trials within 3 months.
14. History of other malignancies within the past 5 years or concurrent other malignancies.
15. Any other condition deemed by the investigator as unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
hPFS | From date of randomization until the date of first documented intrahepatic progression or date of death from any cause, whichever comes first, assessed up to 12 months.
  Intrahepatic Progression-Free Survival (hPFS) assessed by RECIST 1.1

SECONDARY OUTCOMES:
ORR | From date of randomization until the first documented objective response (CR or PR), assessed up to 12 months.
  Objective Response Rate (ORR) assessed by RECIST 1.1
OS | From date of randomization until date of death from any cause, assessed up to 12 months.
  Overall Survival (OS)
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
  Progression-Free Survival (PFS) assessed by RECIST 1.1
DCR | From date of randomization until the first documented objective response (CR or PR) or stable disease (SD), assessed up to 12 months.
  Disease Control Rate (DCR) assessed by RECIST 1.1
MAE | From the time of the baseline procedure (ablation surgery) through 30 days post-procedure
  Incidence of Device-Related Composite Major Adverse Events (MAE)
SAEs | From date of randomization until the end of study visit at 12 months.
  Incidence of All Adverse Events (AEs) and Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital Affiliated to Southeast University, Department of Interventional and Vascular Surgery, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shi DD, Guo JA, Hoffman HI, Su J, Mino-Kenudson M, Barth JL, Schenkel JM, Loeffler JS, Shih HA, Hong TS, Wo JY, Aguirre AJ, Jacks T, Zheng L, Wen PY, Wang TC, Hwang WL. Therapeutic avenues for cancer neuroscience: translational frontiers and clinical opportunities. Lancet Oncol. 2022 Feb;23(2):e62-e74. doi: 10.1016/S1470-2045(21)00596-9. PMID 35114133
- [Background] Chang A, Botteri E, Gillis RD, Lofling L, Le CP, Ziegler AI, Chung NC, Rowe MC, Fabb SA, Hartley BJ, Nowell CJ, Kurozumi S, Gandini S, Munzone E, Montagna E, Eikelis N, Phillips SE, Honda C, Masuda K, Katayama A, Oyama T, Cole SW, Lambert GW, Walker AK, Sloan EK. Beta-blockade enhances anthracycline control of metastasis in triple-negative breast cancer. Sci Transl Med. 2023 Apr 26;15(693):eadf1147. doi: 10.1126/scitranslmed.adf1147. Epub 2023 Apr 26. PMID 37099632
- [Background] Mancusi R, Monje M. The neuroscience of cancer. Nature. 2023 Jun;618(7965):467-479. doi: 10.1038/s41586-023-05968-y. Epub 2023 Jun 14. PMID 37316719
- [Background] Silverman DA, Martinez VK, Dougherty PM, Myers JN, Calin GA, Amit M. Cancer-Associated Neurogenesis and Nerve-Cancer Cross-talk. Cancer Res. 2021 Mar 15;81(6):1431-1440. doi: 10.1158/0008-5472.CAN-20-2793. Epub 2020 Dec 17. PMID 33334813
- [Background] Miller BM, Oderberg IM, Goessling W. Hepatic Nervous System in Development, Regeneration, and Disease. Hepatology. 2021 Dec;74(6):3513-3522. doi: 10.1002/hep.32055. Epub 2021 Aug 15. PMID 34256416
- [Background] Fu Y, Shen K, Wang H, Wang S, Wang X, Zhu L, Zheng Y, Zou T, Ci H, Dong Q, Qin LX. Alpha5 nicotine acetylcholine receptor subunit promotes intrahepatic cholangiocarcinoma metastasis. Signal Transduct Target Ther. 2024 Mar 8;9(1):63. doi: 10.1038/s41392-024-01761-z. PMID 38453934
- [Background] Cui Q, Jiang D, Zhang Y, Chen C. The tumor-nerve circuit in breast cancer. Cancer Metastasis Rev. 2023 Jun;42(2):543-574. doi: 10.1007/s10555-023-10095-1. Epub 2023 Mar 31. PMID 36997828
- [Background] Globig AM, Zhao S, Roginsky J, Maltez VI, Guiza J, Avina-Ochoa N, Heeg M, Araujo Hoffmann F, Chaudhary O, Wang J, Senturk G, Chen D, O'Connor C, Pfaff S, Germain RN, Schalper KA, Emu B, Kaech SM. The beta1-adrenergic receptor links sympathetic nerves to T cell exhaustion. Nature. 2023 Oct;622(7982):383-392. doi: 10.1038/s41586-023-06568-6. Epub 2023 Sep 20. PMID 37731001
- [Background] Mohammadpour H, MacDonald CR, McCarthy PL, Abrams SI, Repasky EA. beta2-adrenergic receptor signaling regulates metabolic pathways critical to myeloid-derived suppressor cell function within the TME. Cell Rep. 2021 Oct 26;37(4):109883. doi: 10.1016/j.celrep.2021.109883. PMID 34706232
- [Background] Huang Q, Hu B, Zhang P, Yuan Y, Yue S, Chen X, Liang J, Tang Z, Zhang B. Neuroscience of cancer: unraveling the complex interplay between the nervous system, the tumor and the tumor immune microenvironment. Mol Cancer. 2025 Jan 17;24(1):24. doi: 10.1186/s12943-024-02219-0. PMID 39825376
- [Background] Vermeer PD, Restaino AC, Barr JL, Yaniv D, Amit M. Nerves at Play: The Peripheral Nervous System in Extracranial Malignancies. Cancer Discov. 2025 Jan 13;15(1):52-68. doi: 10.1158/2159-8290.CD-23-0397. PMID 39801235
- [Background] Zahalka AH, Frenette PS. Nerves in cancer. Nat Rev Cancer. 2020 Mar;20(3):143-157. doi: 10.1038/s41568-019-0237-2. Epub 2020 Jan 23. PMID 31974491
- [Background] Zhang Y, Liao Q, Wen X, Fan J, Yuan T, Tong X, Jia R, Chai P, Fan X. Hijacking of the nervous system in cancer: mechanism and therapeutic targets. Mol Cancer. 2025 Feb 6;24(1):44. doi: 10.1186/s12943-025-02246-5. PMID 39915765
- [Background] Winkler F, Venkatesh HS, Amit M, Batchelor T, Demir IE, Deneen B, Gutmann DH, Hervey-Jumper S, Kuner T, Mabbott D, Platten M, Rolls A, Sloan EK, Wang TC, Wick W, Venkataramani V, Monje M. Cancer neuroscience: State of the field, emerging directions. Cell. 2023 Apr 13;186(8):1689-1707. doi: 10.1016/j.cell.2023.02.002. PMID 37059069